CLINICAL TRIAL: NCT03059589
Title: National Registry of Food Allergy Treatment
Brief Title: Registry of Food Allergy Oral Immunotherapy Treatment
Status: Completed | Type: Observational
Sponsor: Food Allergy Support Team (Other)
Responsible Party: Sponsor
Other Study IDs: Mylan-16-004
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Food Allergy
Keywords: food anaphylaxis; peanut anaphylaxis; food oral immunotherapy; food allergy; food allergy treatment
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this patient registry is to demonstrate safety and efficacy of food oral immunotherapy in food allergic patients. Factors that lead to adverse reactions will be identified. The frequency of rescue epinephrine use will be recorded.

DETAILED DESCRIPTION:
Each participating US clinic is assigned a site number and patients starting food oral immunotherapy will be given a four digit number starting at 0001 within each site. All data will be collected and reported electronically at each clinical site.

ELIGIBILITY:
Inclusion Criteria:

* a history of an allergic reaction following exposure to the food and positive in-vivo or in-vitro sensitivity testing to the food,
* no prior exposure to the food, but markedly high in-vitro specific immunoglobulin E (IgE) to the food

Exclusion Criteria:

* pregnancy
* severe asthma
* poorly controlled atopic dermatitis
* eosinophilic esophagitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to participating clinical sites with high probability of food allergy who choose to undergo food oral immunotherapy treatment.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
efficacy of food allergy treatment | 3 years
  the percentage of patients who successfully reach the maintenance dose of food

SECONDARY OUTCOMES:
epinephrine use | 3 years
  The frequency of epinephrine use during the course of oral immunotherapy as reported in the prospective database. Also, identify factors that are associated with the need for epinephrine.
factors associated with the failure to reach the target dose of food ingestion | 3 years
  Identify factors that are associated with treatment failures through analysis of patient demographics, baseline laboratory test results, and concomitant atopic conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Windom, MD, Principal Investigator
Locations (1):
- Food Allergy Center of FL, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wasserman RL, Factor JM, Baker JW, Mansfield LE, Katz Y, Hague AR, Paul MM, Sugerman RW, Lee JO, Lester MR, Mendelson LM, Nacshon L, Levy MB, Goldberg MR, Elizur A. Oral immunotherapy for peanut allergy: multipractice experience with epinephrine-treated reactions. J Allergy Clin Immunol Pract. 2014 Jan-Feb;2(1):91-6. doi: 10.1016/j.jaip.2013.10.001. PMID 24565775
- [Background] Nachshon L, Goldberg MR, Elizur A, Levy MB, Schwartz N, Katz Y. A Web site-based reporting system for monitoring home treatment during oral immunotherapy for food allergy. Ann Allergy Asthma Immunol. 2015 Jun;114(6):510-5. doi: 10.1016/j.anai.2015.04.007. Epub 2015 May 1. PMID 25940735